CLINICAL TRIAL: NCT03500263
Title: A Phase 1 / 2, Randomized, Double-Blind, Placebo-Controlled Study Designed to Evaluate the Safety, Tolerability, and Pharmacokinetics of PTI-808, PTI-801, and PTI-428 Combination Therapy in Subjects With Cystic Fibrosis
Brief Title: Safety, Tolerability, and Pharmacokinetics of PTI-808, PTI-801, and PTI-428 Combination Therapy in Subjects With Cystic Fibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proteostasis Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PTI-808-02
Record Dates: First submitted 2018-04-09; First posted 2018-04-18 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohorts 1 and 2: PTI-808 Active Co-admin with PTI-801 Active (Active Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 or placebos once-a-day for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: PTI-808; Drug: PTI-801
- Cohorts 1 and 2: PTI-808 Placebo Co-admin with PTI-801 Placebo (Placebo Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 or placebos once-a-day for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: Placebo
- Cohort 3 PTI-808 Active + PTI-801 Active + PTI-428 Active (Active Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 and PTI-428 or placebos once-a-day for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: PTI-808; Drug: PTI-801; Drug: PTI-428
- Cohort 3 PTI-808 placebo + PTI-801 Placebo + PTI-428 Placebo (Placebo Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 and PTI-428 or placebos once-a-day for a total of 14 days. A follow up visit will occur on Day 21.
  Interventions: Drug: Placebo
- Cohort 4 PTI-808 Active + PTI-801 Active + PTI-428 Active (Active Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 and PTI-428 or placebos once-a-day for 7 days immediately followed by PTI-808 co-administered with PTI-801 or placebos once-a-day for 7 days. A follow-up visit will occur on Day 21.
  Interventions: Drug: PTI-808; Drug: PTI-801; Drug: PTI-428
- Cohort 4 PTI-808 Placebo + PTI-801 Placebo + PTI-428 Placebo (Placebo Comparator): Subjects will be randomized to receive either PTI-808 co-administered with PTI-801 and PTI-428 or placebos once-a-day for 7 days immediately followed by PTI-808 co-administered with PTI-801 or placebos once-a-day for 7 days. A follow-up visit will occur on Day 21.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PTI-808 — Active
  Arms: Cohort 3 PTI-808 Active + PTI-801 Active + PTI-428 Active; Cohort 4 PTI-808 Active + PTI-801 Active + PTI-428 Active; Cohorts 1 and 2: PTI-808 Active Co-admin with PTI-801 Active
Drug: Placebo — Placebo
  Arms: Cohort 3 PTI-808 placebo + PTI-801 Placebo + PTI-428 Placebo; Cohort 4 PTI-808 Placebo + PTI-801 Placebo + PTI-428 Placebo; Cohorts 1 and 2: PTI-808 Placebo Co-admin with PTI-801 Placebo
Drug: PTI-801 — Active
  Arms: Cohort 3 PTI-808 Active + PTI-801 Active + PTI-428 Active; Cohort 4 PTI-808 Active + PTI-801 Active + PTI-428 Active; Cohorts 1 and 2: PTI-808 Active Co-admin with PTI-801 Active
Drug: PTI-428 — Active
  Arms: Cohort 3 PTI-808 Active + PTI-801 Active + PTI-428 Active; Cohort 4 PTI-808 Active + PTI-801 Active + PTI-428 Active
Drug: Placebo — Placebo
  Arms: Cohort 3 PTI-808 placebo + PTI-801 Placebo + PTI-428 Placebo; Cohort 4 PTI-808 Placebo + PTI-801 Placebo + PTI-428 Placebo

SUMMARY:
The study is a randomized, double-blind, placebo-controlled, study that will be conducted at multiple centers in subjects with Cystic Fibrosis (CF) who are either homozygous for the F508del mutation or heterozygous with at least copy of the F508del mutation.

DETAILED DESCRIPTION:
Study PTI-808-02 will enroll up to approximately 32 subjects. Subjects in the first cohort will receive PTI-808 and PTI-801. Following completion of Cohort 1, initiation of enrollment into subsequent cohorts will be based upon review and approval by the Safety Review Committee (SRC).

ELIGIBILITY:
Inclusion Criteria:

* Cohorts 1,2 and 4: A Confirmed diagnosis of CF with the F508del/F508del CFTR genotype on record, along with clinical findings consistent with CF such as chronic sinopulmonary disease or gastrointestinal/nutritional abnormalities
* Cohort 3 only: Confirmed diagnosis of CF with at least one copy of the F508del CFTR mutation on record, along with clinical findings consistent with CF, such as chronic sinopulmonary disease or gastrointestinal / nutritional abnormalities
* Forced expiratory volume in 1 second (FEV1) 40-90% predicted, inclusive
* Non-smoker and non-tobacco user for a minimum of 30 days prior to screening
* Cohort 3 only: A sweat chloride value of ≥60 mmol/L based on quantitative pilocarpine iontophoresis (as documented in the subject's medical record or as confirmed at the screening visit)

Exclusion Criteria:

* Currently taking or has taken a CFTR modulator within 30 days prior to initial dose of study drugs
* Participation in another clinical trial or treatment with an investigational agent within 28 days or 5 half-lives, whichever is longer, prior to Study Day 1
* History of cancer within the past 5 years
* History of organ transplantation
* Hospitalization, sinopulmonary infection, CF exacerbation, or other clinically significant infection or illness (as determined by the investigator) requiring an increase or addition of medication, such as antibiotics or corticosteroids, within 14 days of Day 1
* Initiation of any new chronic therapy (e.g., ibuprofen, hypertonic saline, azithromycin, Pulmozyme®, Cayston®, TOBI®) or any change in chronic therapy (excluding pancreatic enzyme replacement therapy) within 28 days prior to Day 1
* History or current evidence of alcohol or drug abuse or dependence within 12 months of screening as determined by the investigator
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measured by the number of subjects who experience adverse events and potentially significant clinical laboratory assessments, electrocardiography, physical examinations, vital signs. | Baseline through Day 21

SECONDARY OUTCOMES:
Apparent terminal half-life (t1/2) of multiple oral doses of PTI-808 + PTI-801 and PTI-428 (cohorts 3 & 4 only) | Day 1 through 15
Time to reach maximum plasma concentration (Tmax) of multiple oral doses of PTI-808 + PTI-801 and PTI-428 (cohorts 3 & 4 only) | Day 1 through 15
Maximum plasma concentration (Cmax) of multiple oral doses of PTI-808 + PTI-801 and PTI-428 (cohorts 3 & 4 only) | Day 1 through 15
Change in FEV1 over time | Baseline through Day 21

OTHER OUTCOMES:
Change in sweat chloride over time | Baseline through Day 21
Change in weight over time | Baseline through Day 21
Change in BMI over time | Baseline through Day 21
Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) respiratory domain results over time | Baseline through Day 21
  Disease-specific instrument designed to measure impact on overall health, daily life, perceived well-being and symptoms. Developed specifically for use in patients with a diagnosis of cystic fibrosis.
  Scaling of items:
  5 distinct 4-point Likert scales (e.g., always/often/ sometime/never)
  Scoring:
  Scores for each HRQoL domain; after recoding, each item is summed to generate a domain score and standardized. Scores range from 0 to 100, with higher scores indicating better health.
Change in nasal epithelial mRNA expression over time | Baseline through Day 21
Change in nasal protein expression over time | Baseline through Day 21

CONTACTS AND LOCATIONS:
Locations (4):
- United Kingdom (4):
  - Celerion, Belfast
  - Western General Hospital, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Medicines Evaluation Unit, Manchester

IPD SHARING:
Plan to Share IPD: Yes